CLINICAL TRIAL: NCT05560399
Title: A Multicenter Phase 1-DEC (Dose Expansion Cohort) Open-label Study of Iberdomide (CC-220) in Combination With Elotuzumab and Dexamethasone for Relapsed/Refractory Multiple Myeloma
Brief Title: A Study of Iberdomide (CC-220) in Combination With Elotuzumab and Dexamethasone for Relapsed/Refractory Multiple Myeloma
Acronym: CC-220
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Multiple Myeloma Research Consortium (Network); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Cesar Rodriguez Valdes, Associate Professor of Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCO 22-0016
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — iberdomide; elotuzumab; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Part 1 is a dose-finding evaluation of Iberdomide in combination with Elotuzumab and Dexamethasone at their approved doses for patients with relapsed/refractory multiple myeloma.
  Part 2 of this study is an open-label, single-arm dose expansion cohort that will enroll additional patients at the recommended maximum tolerated dose of Iberdomide as determined in Part 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Iberdomide, Elotuzumab and Dexamethasone (Experimental): Dose-Finding: Patients will be enrolled in a 3+3 dose escalation cohort. Dose-Expansion: additionally enrolled patients at the recommended maximum tolerated dose of Iberdomide as was determined in Part 1 (Dose-Finding Phase).
  Interventions: Drug: Iberdomide; Drug: Elotuzumab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Iberdomide — Route of administration: oral pill. Schedule: Taken Once daily on days 1-21. Dose: will be tested at 1 mg, 1.3 mg, and 1.6mg. 1mg dose may be reduced to 0.75mg if not tolerated.
  Other Names: CC-220
Drug: Elotuzumab — Route of administration: IV Dose: 10 mg/kg for cycles 1 and 2. 20 mg/kg for cycle 3 and beyond. Schedule: Days 1, 8, 15, and 22 for cycles 1 and 2. Then taken on Day 1 (every 28 days) of each cycle thereafter.
Drug: Dexamethasone — Route of administration: Oral pill or IV Dose: 36 mg within 24 hrs of day 1 of each cycle and day 8, 15, and 22 of cycle 1 and 2.
  40 mg on days 8, 15, 22 of cycle 3 and all subsequent cycles. (20 mg for > 75 years old).
  Schedule: On days that Elotuzumab is administered, Dexamethasone to be taken 28mg orally (for ≤75 years old) or 8mg orally (for > 75 years old) between 3 and 24 hours before Elotuzumab plus 8 mg IV between 45 and 90 minutes before Elotuzumab for all patients.
  On days that Elotuzumab is not administered but a dose of Dexamethasone is scheduled (Days 8, 15, and 22 of cycle 3 and all subsequent cycles), 40 mg orally for ≤75 years older and 20 mg for

SUMMARY:
This is a single-arm, open-label study evaluating the safety, tolerability and efficacy of Iberdomide (CC-220) in combination with Elotuzumab and Dexamethasone in patients with RRMM. The researchers hypothesize that the combination of Iberdomide and Elotuzumab will synergize to promote myeloma cell death, resulting in an overall response rate of at least 53%, with an acceptable safety profile. Patients will be enrolled in a 3+3 dose escalation cohort to evaluate the safety of this combination and to establish the MTD (maximum tolerated dose). The MTD will be the dose for the patients enrolled in dose expansion cohort. A total maximum of 37 patients will be recruited: maximum 18 patients will be recruited in the dose escalation phase, followed by an additional 19 patients in the dose expansion cohort for a total of 25 patients treated at the MTD.

DETAILED DESCRIPTION:
Part 1 is an open-label, sequential allocation, dose-finding evaluation of the sequential administration of Iberdomide in combination with Elotuzumab and Dexamethasone at their approved doses for patients with relapsed/refractory multiple myeloma. This phase will follow a standard 3+3 design. During this phase, the maximum tolerated dose of Iberdomide in combination with Elotuzumab and Dexamethasone will be determined and recommended for the dose expansion cohort.

Part 2 of this study is an open-label, single-arm dose expansion cohort that will enroll additional patients at the recommended maximum tolerated dose of Iberdomide as determined in Part 1. Researchers will continue to verify the safety and tolerability of this combination and examine the anti-myeloma activity of the regimen. In addition to measuring overall response rate, duration of response, and survival data, researchers will explore the effect of this combination on the biology of multiple myeloma and the immune system in order to gain insight into patterns of response that may help predict patient population most-likely to benefit from this treatment in the future.

ELIGIBILITY:
Inclusion Criteria

* Subject is ≥18 years of age at the time of signing the informed consent form (ICF).
* Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
* Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
* All subjects must have documented diagnosis of MM with disease progression per IMWG criteria during or after their last anti-myeloma therapy (Appendix D).
* All subjects must have measurable disease at screening, defined as one or more of the following:

  1. Serum IgG, IgA, IgM M-protein ≥ 0.5 g/dL
  2. Urinary M-Protein ≥ 200 mg urinary M-protein excretion in a 24-hour collection sample
  3. Involved serum free light chain (sFLC) ≥ 10 mg/dL provided the FLC ratio is abnormal.
* All patients must have ECOG Performance Status ≤ 2 (Appendix A).
* Subjects must have received at least 1 and at most 3 lines of therapy (note: induction and stem cell transplants with or without maintenance therapy is considered 1 line of therapy) including at least one IMiD (thalidomide, lenalidomide, pomalidomide), a proteosome inhibitor (bortezomib, carfilzomib, ixazomib), and an anti-CD38 agent (daratumumab, isatuximab).
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy tests (minimum sensitivity 25 IU/L or equivalent units of HCG), at 10-14 days prior to start of study drug; another within 24 hours prior to the start of study drug.
* Women must not be breastfeeding
* WOCBP must agree to follow instructions for method(s) of contraception for 1 month (4 weeks) before the start of treatment with study drugs, for the duration of treatment with study drugs, and for a total of 5 months post-treatment completion. This includes 2 methods of reliable birth control simultaneously:

  1. one highly effective form of contraception - tubal ligation, IUD, hormonal (birth control pills, injections, hormonal patches, vaginal rings, or implants), or partner's vasectomy, and;
  2. additional effective contraceptive method - male latex or synthetic condom, diaphragm, or cervical cap. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy.
* Males who are sexually active with WOCBP must always use a latex or synthetic condom during any sexual contact with females of reproductive potential while taking Iberdomide (CC-220) and for up to 90 days after discontinuing Iberdomide (CC-220), even if they have undergone a successful vasectomy. Male patients must not donate sperm.
* Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, they must still undergo pregnancy testing as described in this section.
* All subjects must agree not to share study medication.
* Male subjects receiving Elotuzumab must agree to follow instructions for method(s) of contraception for 1 month (4 weeks) before the start of treatment with study drugs, for the duration of treatment with study drugs, and for a total of 7 months post treatment completion.
* Subjects must be willing to refrain from blood donations during study drug therapy and for 90 days after therapy.

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

* Subjects with solitary bone or extramedullary plasmacytoma as the only evidence of plasma cells dyscrasia.
* Subjects with monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), primary amyloidosis (no active multiple myeloma), Waldenström's macroglobulinemia, or POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Subjects with active plasma cell leukemia (defined as either 20% of peripheral blood white blood cell count comprised of plasma/CD138+ cells or an absolute plasma cell count of 2 x 109/L)
* Subjects with Central Nervous System involvement with multiple myeloma
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the informed consent form
* Any serious concurrent medical conditions that may make the patient non-evaluable or put the patient's safety at risk
* Active infection that requires parenteral anti-infective treatment >14 days
* Unable to tolerate thromboembolic prophylaxis while on the study
* Severe hypersensitivity reaction to prior IMiD (thalidomide, lenalidomide or pomalidomide)
* Grade > 2 peripheral neuropathy (per NCI CTCAE v5.0)
* Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection.
* Known HIV infection or known acquired immunodeficiency syndrome (AIDS).
* Prior or concurrent malignancy, except for the following:

  1. Adequately treated basal cell or squamous cell skin cancer or in-situ carcinoma.
  2. Any other cancer from which the subject has been disease free for > 3 years prior to study entry.
* Prior treatment with Iberdomide (CC-220)
* Prior treatment with Elotuzumab
* Use of any anti-myeloma drug therapy within 14 days of the initiation of study drug treatment or use of any experimental drug therapy within 28 days of the initiation of study drug treatment
* Treatment with melphalan within 4 weeks of the first dose of study drug
* Treatment with corticosteroids (other than the Dexamethasone of anti-myeloma regimens) within 3 weeks of the first dose of study drug, except for the equivalent of ≤ 10 mg prednisone per day or corticosteroids with minimal to no systemic absorption (i.e., topical or inhaled corticosteroids)
* Prior autologous stem cell transplant within 12 weeks of the first dose of study drug
* Prior allogeneic stem cell transplant except subjects who have completed the stem cell transplant > 12 months prior to first dose of study drug, have no history of graft versus host disease, and are not on systemic immunosuppressive therapy
* Major cardiac surgery within 8 weeks prior to the first dose of study drug; all other major surgery within 4 weeks prior to the first dose of study drug.
* Subjects with following physical and laboratory test findings:

  1. Absolute neutrophil count < 1 x 109/L without growth factor support within 1 week
  2. Platelets < 75 x 109/L without transfusion support within 3 days for the dose escalation phase. For the DEC: platelets < 75 x 109/L or < 30 x 109/L if ≥ 50% of bone marrow nucleated cells were plasma cells without transfusion support within 3 days
  3. Hemoglobin < 8 g/dL without transfusion support within 3 days of screening
  4. Creatinine clearance < 30 ml/min according to the Cockroft-Gault formula:

     * Female CrCl = [(140 - age in years) x weight in kg x 0.85] / [72 x serum creatinine in mg/dl]
     * Male CrCl = [(140 - age in years) x weight in kg x 1.00] / [72 x serum creatinine in mg/dl]
  5. Total bilirubin ≥ 2 x ULN (≥ 3 x ULN if documented Gilbert's syndrome)
  6. AST or ALT ≥ 3x ULN
  7. Corrected serum calcium > 13.5 mg/dL
* Subjects with known severe hypersensitivity or anaphylaxis to Dexamethasone, any excipients in Elotuzumab, formulation or recombinant protein, or any monoclonal antibody
* Use of strong CYP3A inhibitors within 2 weeks or 5 half-lives of the drug whichever is shorter prior to the first dose of study drug during the dose escalation portion of the study. (In the dose expansion part, strong CYP3A inhibitors may be allowed with appropriate dose adjustments based on the results of the itraconazole drug-drug interaction study. The concomitant use of strong CYP3A induces should be avoided.)
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Iberdomide dose limiting toxicity | 28 days
  The dose limiting toxicity (DLT) rate at the Maximum Tolerated Dose, defined as the proportion of patients in the safety population of the study that experience at least 1 DLT within the first cycle of Iberdomide (CC-220) in combination with Elotuzumab and Dexamethasone treated at the maximum tolerated dose (MTD).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to 3 months
  Overall Response Rate (ORR) is defined as the proportion of patients treated at the MTD of Iberdomide (CC-220) in combination with Elotuzumab and Dexamethasone in both phase 1 and DEC phase of the study that achieved best overall response of PR or better (Stringent Complete Response (sCR); Complete Response (CR); Very good partial response (VGPR); Partial Response (PR), according to International Myeloma Working Group (IMWG) criteria at Cycle 4 Day 1 (C4D1).
Number of adverse events (AE) | up to 3 months
  Number of Adverse Events (AE) - an AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure
Progression-free survival (PFS) | up to 3 months
  PFS: is defined as the duration of time from start of treatment to the first occurrence of disease progression or death on study from any cause, whichever occurs earlier
Best Overall Response Rate (BOR) | up to 3 months
  Best Overall Response Rate (BOR) is defined as the proportion of patients treated at the MTD of Iberdomide (CC-220) in combination with Elotuzumab and Dexamethasone in both phase 1 and DEC phase of the study that achieved sCR, CR, VGPR, PR, minimal response, and Stable Disease (SD), according to IMWG criteria at any evaluation assessment prior to progression of disease as their best response.
Duration of Response (DOR) | up to 3 months
  Duration of Response (DOR) is defined as the time from achieving a PR or better to progression, per 2016 IMWG criteria
Overall Survival (OS) | up to 3 months
  Overall survival is defined from time from initiation of treatment to death by any cause
Clinical Benefit Rate | up to 3 months
  Clinical Benefit Rate is the proportion of patients treated at the MTD of Iberdomide (CC-220) in combination with Elotuzumab and Dexamethasone in both phase 1 and DEC phase of the study that achieved best overall response of minimal response or better (sCR + CR + VGPR + PR + minimal response [MR]) according to the IMWG criteria at C4D1
Disease Control Rate | up to 3 months
  Disease Control Rate is the proportion of patients treated at the MTD of Iberdomide (CC-220) in combination with Elotuzumab and Dexamethasone in both phase 1 and DEC phase of the study that achieved best overall response of stable disease or better (sCR + CR + VGPR + PR + MR + SD) according to the IMWG criteria at C4D1

CONTACTS AND LOCATIONS:
Overall Officials: Samir Parekh, MBBS, Principal Investigator — Icahn school of medicine; Cesar Rodriguez, MD, Study Chair — Icahn School of Medicine
Locations (1):
- Icahn School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

DOCUMENTS (1):
  • Informed Consent Form (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT05560399/ICF_000.pdf